CLINICAL TRIAL: NCT06341712
Title: A Phase II, Randomized, Open-label Study to Assess the Efficacy, Safety, and Pharmacokinetics (PK) of Maintenance Cabozantinib (XL184) Plus Best Supportive Care (BSC) Versus BSC in Children, Adolescents and Young Adults (AYA) With Unresectable Residual Osteosarcoma Either at Diagnosis or at First Relapse After Standard Treatment
Brief Title: Effects of Maintenance Cabozantinib+BSC Versus BSC in Children and AYA With Osteosarcoma
Acronym: CabOSTar
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-60000-461; 2023-506229-12-00 (Other: Ipsen)
Record Dates: First submitted 2024-03-04; First posted 2024-04-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma; Osteosarcoma in Children; Osteosarcoma in Adolescents and Young Adults
Keywords: Osteosarcoma; Cabozantinib; Children; Osteosarcoma in adolescents and young adults (AYA); AYA
MeSH Terms: conditions — Osteosarcoma | interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Cabozantinib+ Best supportive care (BSC) (Experimental): Participants will receive cabozantinib and BSC.
  Interventions: Drug: Cabozantinib; Other: Best Supportive Care (BSC)
- Arm B: Best supportive care (BSC) (Other): Participants will receive BSC alone administered per investigator's discretion and institutional guidelines.
  Interventions: Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Cabozantinib — Participants will receive cabozantinib orally Once daily (QD) on a continuous dosing schedule for cycles of 28 days.
  Arms: Arm A: Cabozantinib+ Best supportive care (BSC)
Other: Best Supportive Care (BSC) — Participants will receive BSC. BSC includes antibiotics, nutritional support, correction of metabolic disorders, optimal symptom control and pain management (including palliative radiotherapy), etc. but does not include tumor specific therapy.
  Arms: Arm A: Cabozantinib+ Best supportive care (BSC)
Other: Best Supportive Care (BSC) — Participants will receive BSC alone. BSC includes antibiotics, nutritional support, correction of metabolic disorders, optimal symptom control and pain management (including palliative radiotherapy), etc. but does not include tumor specific therapy.
  Arms: Arm B: Best supportive care (BSC)

SUMMARY:
The participants of this study will be children, adolescents, and young adults with residual osteosarcoma, which cannot be removed completely through surgery.

Participants will have achieved a partial response or stable disease at the end of conventional chemotherapy. Osteosarcoma is cancer of the bone. The cancer cells make immature bone cells, known as osteoid.

Osteosarcoma is very rare, but it is the most common type of bone cancer in children and teens. It is most common in teens and young adults.

In this study, participants will receive either cabozantinib and best supportive care or the best supportive care alone. Best supportive care will be provided at the investigator's discretion and according to institutional guidelines.

It includes antibiotics, nutritional support, correction of metabolic disorders, optimal symptom control and pain management (including radiotherapy), etc. but does not include tumor specific therapy.

Cabozantinib will be taken by mouth (orally), as a tablet, once a day. Cabozantinib will be provided to participants who tolerate it for as long as their disease does not progress. Participants in the study receiving best supportive care alone may switch to treatment with cabozantinib and best supportive care if their disease progresses and if other eligibility criteria are met.

Participants may withdraw consent to participate at any time.

The estimated duration of the study for participants is 24 months, however a participant could remain in the study longer if demonstrating treatment benefit.

ELIGIBILITY:
Inclusion Criteria :

* Participants must be ≥5 and ≤30 years of age at the time of study entry.
* Histologically or cytologically confirmed diagnosis of high-grade osteosarcoma as defined by a local pathologist
* Participants with unresectable residual disease after standard chemotherapy treatment at diagnosis or first relapse (treated with systemic chemotherapy). A minimum of 4 cycles of systemic chemotherapy (or minimum of 2 cycles if chemotherapy was stopped early due to toxicity) must have been received.
* Measurable residual or evaluable disease by RECIST version 1.1. Participants will be considered with evaluable disease if they have only non-measurable disease as per RECIST version 1.1 criteria.
* Absence of Progressive Disease (PD) (defined by the investigator according to RECIST version 1.1) at study entry. Note, the two most recent radiological evaluations (e.g. computerised tomography (CT) or magnetic resonance resonance imaging (MRI) scan) including the one following completion of chemotherapy should be available later to facilitate BIRC review.
* Chemotherapy must be the last anticancer treatment received by participants before study entry and must have been completed at least 4 weeks but no longer than 2 months before randomization.
* Participants must have recovered to Grade ≤1, except for alopecia, ototoxicity, and Grade ≤2 peripheral neuropathy, per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) from the acute toxic effects of all prior anticancer therapy at study entry, unless AEs are clinically non significant and/or stable on supportive therapy, per investigator clinical judgment.
* Life expectancy >6 months.
* Performance level: participants must have a Lansky or Karnofsky performance status score of ≥70 corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0-1.
* Adequate organ and marrow function.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications.
* Male and/or female (according to their reproductive organs and functions assigned by chromosomal complement) (FDA 2016)
* Contraception and barriers as well as pregnancy testing is required as appropriate for the age and sexual activity of pediatric participants and as required by local regulations.
* All participants (typically ≥18 years) and/or their parents or legal guardians must sign a written informed consent and assent must be obtained from minor participants according to local guidelines.

Exclusion Criteria :

* Low grade osteosarcoma and periosteal osteosarcoma
* Previous treatment with cabozantinib or another Mesenchymal-epithelial transition (MET)/hepatocyte growth factor (HGF) inhibitor (e.g., tivantinib, crizotinib).
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks or 5 half-lives of the agent, whichever is longer, before first dose of study intervention.
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study intervention (or washout of at least 5 half-lives, whichever is shorter).
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery or major surgery e.g., removal or biopsy of brain metastasis) and stable for at least 4 weeks prior to randomization. Eligible participants must be neurologically asymptomatic and without systemic corticosteroid treatment at the time of randomization. Note: Participants with a known seizure disorder who are receiving non-enzyme inducing anticonvulsants and have well-controlled seizures on a stable dose of anti-convulsant may be enrolled.
* Participants who have an uncontrolled/active infection requiring systemic therapy.
* Participants who are unable to swallow intact tablets.
* Participants with uncontrolled, significant intercurrent or recent illness.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Any other active malignancy at time of first dose of study intervention or diagnosis of another malignancy within 3 years prior to first dose of study intervention that requires active treatment.
* Pregnancy or breast-feeding.
* Participants who in the opinion of the investigator may not be able to comply with the requirements of the study are not eligible
* Major surgery (eg, orthopaedic surgery, removal or biopsy of brain metastasis) within 8 weeks before randomization. Complete wound healing from major surgery must have occurred 4 weeks before randomization and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before randomization. Participants with clinically relevant ongoing complications from prior surgery are not eligible.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) assessed by Blinded Independent Radiology Committee (BIRC) | From randomization until disease progression or death from any cause, whichever occurs first (approximately 34 months).
  PFS defined as the time from the date of randomization to the date of first documented disease progression or the date of death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate assessed by BIRC | 4 months and 1 year after randomization.
  PFS rate at 4 months and 1 year was defined as the probability that participants have not progressed by BIRC assessment and remain alive at 4 months and 1 year.
Objective response rate (ORR) assessed by BIRC | Approximately 34 months after randomization.
  ORR defined as the proportion of participants who have achieved complete response (CR) or partial response (PR) determined by BIRC.
Disease control rate (DCR) assessed by BIRC | Approximately 34 months after randomization.
  Defined as the proportion of participants who have achieved CR, PR, or stable disease (SD) determined by BIRC
PFS assessed by investigator | From randomization until disease progression or death from any cause, whichever occurs first (approximately 34 months).
  Defined as the time from the date of randomization to the date of first documented disease progression determined by investigator or the date of death due to any cause, whichever occurs first
PFS rate assessed by investigator | At 4 months and 1 year after randomization.
  Defined as the probability that participants have not progressed by investigator assessment and remain alive at 4 months and 1 year.
ORR assessed by investigator | Approximately 34 months after randomization.
  Defined as the proportion of participants who have achieved complete response (CR) or partial response (PR) determined by investigator using RECIST version 1.1.
DCR assessed by investigator | Approximately 34 months after randomization.
  Defined as the proportion of participants who have achieved CR, PR, or SD determined by investigator.
Overall survival (OS) | From randomization until death or last contact (approximately 34 months).
  Defined as the time from date of randomization to the date of death, from any cause
1-year overall survival rate | At 1 year after randomization.
  Defined as the probability participants alive at 1 year.
Percentage of participants with Treatment Emergent Adverse Event (TEAEs) and Adverse Events of Special Interest (AESIs). | From screening to 30 days after last dose.
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Area Under Curve (AUC) at steady state. | At Day 1 of week 1 and Day 1 of week 5.
Average concentration (Cavg) at steady state | At Day 1 of week 1 and Day 1 of week 5.
Minimum concentration (Cmin) at steady state | At Day 1 of week 1 and Day 1 of week 5.
Maximal concentration (Cmax) at steady state | At Day 1 of week 1 and Day 1 of week 5.
Acceptability and palatability in children and adolescents assessed using a horizontal visual assessment scale. | Day of first dose.
  Five-point Facial Hedonic Scale (FHS) with a correlated 100-point horizontal Visual Analog Scale (VAS) (FHS/VAS-5) will be used to assess acceptability and palatability in children and adolescents. Final scores range from 0 to 100, with higher scores indicating better palatability and acceptability.
Change from baseline in score for all Paediatric QoL Inventory (PedsQL) Scales including Generic Core Scales and Cancer Modules. | From screening to 30 days after last dose.
  The PedsQL is a modular instrument designed to measure health-related quality of life in children and adolescent. The PedsQL generic core scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL. The PedsQL cancer modules was designed to measure paediatric cancer specific HRQoL. Final total scores range from 0 to 100, with higher scores indicating better health related quality of life.
Change from baseline in European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) (EORTC QLQ-C30) for adult participants | From screening to 30 days after last dose.
  The EORTC QLQ-C30 was developed by the EORTC Quality of Life Group to assess HRQoL, functioning, and symptoms in cancer clinical trials. It is a 30-item self-administered questionnaire for all cancer types. Final scores range from 0 to 100, with higher scores indicating better health related quality of life. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (16):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States
- University Hospital Gent, Ghent, Belgium
- Canada (2):
  - McGill University Health Centre - Centre for Innovative Medicine, Québec
  - Princess Margaret cancer center, Toronto
- Centre Oscar Lambret, Lille, France
- Germany (2):
  - Universitätsmedizin Mainz, Mainz
  - Dr. von Haunerschen Kinderspital, München
- Italy (2):
  - Ospedale Ortopedico Rizzoli di Bologna, Bologna
  - AOU Città della Salute e della Scienza di Torino, Piemonte
- Amsterdam UMC - Locatie AMC, Amsterdam, Netherlands
- Instytut Matki i Dziecka, Warsaw, Poland
- Spain (4):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/